CLINICAL TRIAL: NCT00282815
Title: Treatment of Obstructive Sleep Apnea After Stroke
Brief Title: Sleep Apnea Treatment After Stroke (SATS)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor recruitment. Funding expired.
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Devin Brown, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: K23NS051202 (NIH)
Record Dates: First submitted 2006-01-26; First posted 2006-01-27 (Estimated); Results first posted 2013-03-11 (Estimated); Last update posted 2013-03-11 (Estimated); Status verified 2012-12

CONDITIONS: Obstructive Sleep Apnea; Stroke
Keywords: obstructive sleep apnea; stroke; OSA; CPAP; continuous positive airway pressure
MeSH Terms: conditions — Sleep Apnea, Obstructive; Stroke | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): CPAP
  Interventions: Device: continuous positive airway pressure or CPAP
- 2 (Sham Comparator): sham CPAP (placebo)
  Interventions: Device: sham CPAP

INTERVENTIONS:
Device: continuous positive airway pressure or CPAP — RemStar Pro (Respironics, Inc.) The CPAP is applied through a nasal mask during the hours of sleep. Positive air pressure holds the naso-oro-pharyngeal airway open during sleep.
  Arms: 1
Device: sham CPAP — sham CPAP
  Arms: 2

SUMMARY:
The purpose of this study is to determine if treating stroke patients who have obstructive sleep apnea with continuous positive airway pressure will improve symptoms caused by the stroke.

DETAILED DESCRIPTION:
Stroke is the leading cause of adult disability in the United States, yet there are very few treatments that improve stroke outcome. Obstructive sleep apnea (OSA)--frequent upper airway blockage that occurs during sleep--is common after stroke, affecting more than half of stroke patients. The most common treatment for obstructive sleep apnea in the general population is nasal continuous positive airway pressure (CPAP) applied through a nasal mask during the hours of sleep. Positive air pressure holds the naso-oro-pharyngeal airway open during sleep.

The objective of this single-center, prospective, randomized study is to evaluate CPAP treatment in post-stroke patients. Participants will go through a medical interview, a brief neurological examination, and a sleep study to screen them for OSA. Those with OSA will be eligible for the second phase of the study during which participants will be randomly selected to receive either treatment with CPAP or with sham CPAP (placebo).

This project promises to establish feasibility, develop design and identify suitable outcome measures (e.g. hours of CPAP treatment per week, functional outcome, depression, fatigue, and impaired alertness) for a large-scale clinical trial of CPAP in stroke patients with OSA. If the larger trial shows benefits of CPAP, a new treatment for more than half of all stroke patients will become available.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke within 7 days of planned polysomnography/sleep screening study
* Modified Rankin Scale score >1
* If of child-bearing potential, has a negative urine or serum pregnancy test

Exclusion Criteria:

* Decompensated heart failure
* Cardiac or respiratory arrest within the past 3 months
* Myocardial infarction within the past 3 months
* Severe pneumonia
* Hypertension refractory to treatment
* Any other unstable medical condition which is thought to interfere with participation
* Known preexisting OSA already on CPAP or previously failed CPAP or used CPAP
* Previous pneumothorax
* Bullous emphysema
* Chronic obstructive pulmonary disease (COPD), obesity-hypoventilation, or another condition warranting the use of nasal bilevel positive airway pressure instead of CPAP
* Acute sinus or ear infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2004-09; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Devin Brown, MD, MS, Principal Investigator — Associate Professor, Stroke Program, University of Michigan; Lewis Morgenstern, MD, Study Director — Director, Stroke Program, University of Michigan; Jack Kalbfleisch, PhD, Study Director — University of Michigan Dept of Biostatistics
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Brown DL, Chervin RD, Kalbfleisch JD, Zupancic MJ, Migda EM, Svatikova A, Concannon M, Martin C, Weatherwax KJ, Morgenstern LB. Sleep apnea treatment after stroke (SATS) trial: is it feasible? J Stroke Cerebrovasc Dis. 2013 Nov;22(8):1216-24. doi: 10.1016/j.jstrokecerebrovasdis.2011.06.010. Epub 2011 Jul 23. PMID 21784661

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled from inpatient neurology service.
Groups:
- Sham Continuous Positive Airway Pressure (CPAP): Subtherapeutic CPAP
Period: Overall Study
Arm/Group | Active Continuous Positive Airway Pressure (CPAP) | Sham Continuous Positive Airway Pressure (CPAP)
Started | 15 | 17
Completed | 8 | 11
Not Completed | 7 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Continuous Positive Airway Pressure (CPAP) | Sham Continuous Positive Airway Pressure (CPAP) | Total
Number analyzed (Participants) | 15 | 17 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 5 | 13
  >=65 years | 7 | 12 | 19
Age Continuous [Mean (Standard Deviation); unit: years] | 61 (16) | 74 (16) | 65 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 4 | 14
  Male | 5 | 13 | 18
Region of Enrollment [Number; unit: participants]
  United States | 15 | 17 | 32

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Continuous Positive Airway Pressure (CPAP)/Sham CPAP Usage Hours Over the 3 Month Period.
Time Frame: 3 months
Population: Data not available on one sham participant (lowering n from 11 to 10 in the shame group).
Measure: Median (Inter-Quartile Range); unit: Hours/participant
Arm/Group | Active CPAP | Sham CPAP
Number analyzed (Participants) | 8 | 10
Hours/participant | 53 [22 to 173] | 74 [17 to 94]

2. Primary Outcome: Number of Subjects Who Withdraw From Study.
Description: Prespecified outcome.
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | After Randomization
Number analyzed (Participants) | 32
participants | 13

3. Secondary Outcome: Barthel Index
Description: Barthel Index score range: 0 (worst, fully dependent) - 100 (best, independent).
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: units on a scale (range 0-100)
Arm/Group | Active Continuous Positive Airway Pressure (CPAP) | Sham Continuous Positive Airway Pressure (CPAP)
Number analyzed (Participants) | 8 | 11
units on a scale (range 0-100) | 95 [90 to 100] | 100 [95 to 100]

ADVERSE EVENTS:
Arm/Group | Active Continuous Positive Airway Pressure (CPAP) | Sham Continuous Positive Airway Pressure (CPAP)
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/17
Other Adverse Events (participants affected / at risk) | 0/15 | 0/17

LIMITATIONS AND CAVEATS:
Attrition pre-randomization and while in randomized treatment led to small numbers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No